CLINICAL TRIAL: NCT01325545
Title: Detection of Occult Paroxysmal Atrial Fibrillation in Patients With Cryptogenic Stroke or TIA Using 21-Day Mobile Cardiac Outpatient Telemetry
Brief Title: Detection of Occult Paroxysmal Atrial Fibrillation After Stroke Using Prolonged Ambulatory Cardiac Monitoring
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Cardionet (Industry)
Responsible Party: Principal Investigator, Alejandro Rabinstein, Professor of Neurology, Mayo Clinic
Other Study IDs: 08-003788
Record Dates: First submitted 2011-03-28; First posted 2011-03-29 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Stroke; Atrial Fibrillation
Keywords: Stroke; Atrial Fibrillation
MeSH Terms: conditions — Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cryptogenic stroke: Patients with stroke of unknown cause after comprehensive conventional evaluation
  Interventions: Other: Mobile cardiac rhythm monitoring
- Stroke of known cause: Patients with stroke of known cause determined by comprehensive conventional evaluation
  Interventions: Other: Mobile cardiac rhythm monitoring

INTERVENTIONS:
Other: Mobile cardiac rhythm monitoring — Continuous ambulatory cardiac rhythm monitoring using the CardioNet MCOT device

SUMMARY:
About one-third of patients with stroke have no documented cause for the cerebrovascular event (known as cryptogenic strokes). Atrial fibrillation is a common cause of stroke, but when transient (paroxysmal) it may remain undiagnosed. Recent data suggest that occult paroxysmal atrial fibrillation may be identified in patients with cryptogenic strokes using prolonged ambulatory cardiac rhythm monitors.

The investigators designed this study pursuing the following goals:

1. To determine the prevalence of occult paroxysmal atrial fibrillation in patients with cryptogenic stroke using long-term mobile cardiac outpatient telemetry.
2. To compare this prevalence to that found in a control group with stroke of known, non-cardioembolic cause.
3. To look for clinical, laboratory, echocardiographic, and imaging data that serve as risk factors for occult paroxysmal atrial fibrillation in patients with cryptogenic stroke.
4. To examine the utility of mobile cardiac outpatient telemetry, a relatively new diagnostic tool, in the evaluation of patients with cryptogenic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Stroke or TIA within previous 3 months
* Stroke work up including: EKG, serum lipids, serum TSH, TTE or TEE, brain CT and/or MRI, Vascular Evaluation of head and neck using any combination of ultrasound, MRA, CTA, and conventional angiography

Exclusion Criteria:

* Documented history of atrial fibrillation or flutter
* PFO closure planned before conclusion of the monitoring period
* Incomplete stroke work up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stroke or TIA confirmed by a vascular neurologist within previous 3 months with complete evaluation for stroke causes according to current standards.
Sampling Method: Non-Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Detection of Atrial Fibrillation | 21 days
  Documented presence of atrial fibrillation detected by the monitoring device and independently confirmed by a board-certified cardiologist

SECONDARY OUTCOMES:
Time to first episode of atrial fibrillation | Within monitoring period (3 weeks)
Atrial Fibrillation Load | Within monitoring period (3 weeks)
  Total time that the patient had atrial fibrillation during the monitoring period
Adverse events related to mobile cardiac monitoring | 21 days
Symptomatic status of episode of atrial fibrillation | 21 days
  Presence or absence of symptoms related to the occurrence of paroxysmal atrial fibrillation
Longest duration of episode of atrial fibrillation | 21 days

REFERENCES:
- [Derived] Baturova MA, Sheldon SH, Carlson J, Brady PA, Lin G, Rabinstein AA, Friedman PA, Platonov PG. Electrocardiographic and Echocardiographic predictors of paroxysmal atrial fibrillation detected after ischemic stroke. BMC Cardiovasc Disord. 2016 Nov 3;16(1):209. doi: 10.1186/s12872-016-0384-2. PMID 27809773